CLINICAL TRIAL: NCT07368257
Title: Replication and Evaluation of the RISE-APS Model In New Contexts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RISE Collaborative (Other)
Collaborators: Ventura County APS (Unknown); Harris County APS (Unknown); Cuyahoga County APS (Unknown); ONEgeneration (Unknown); Harris County AAA (Unknown); Benjamin Rose (Unknown); Northwest District APS (Unknown); West Central Texas AAA (Unknown)
Responsible Party: Principal Investigator, David Burnes, Professor, Director of Research and Evaluation, RISE Collaborative
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90EJIG0055-01-00; 90EJIG0055-01-00 (Other Grant/Funding Number: Administration for Community Living)
Record Dates: First submitted 2025-10-24; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Elder Abuse; Self-Neglect
Keywords: Elder Abuse; Self-Neglect; RISE; Adult Protective Services

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APS Only (Experimental): Participants in this arm will receive usual care Adult Protective Services (APS) on its own.
  Interventions: Behavioral: APS
- RISE-APS (Active Comparator): Participants in this arm will receive both Adult Protective Services (APS) and RISE (Repair Harm, Inspire Change, Support Connection, Empower Choice)
  Interventions: Behavioral: RISE; Behavioral: APS

INTERVENTIONS:
Behavioral: RISE — RISE works with cases involving older adults who are at risk of (prevention) or experiencing (response intervention) OAM. The model operates at Relational, Individual, Social, and Environmental levels and, through its core modalities, the intervention seeks to Repair Harm (restorative approaches), Inspire Change (motivational interviewing), Support Connection (teaming), and Empower Choice (supported decision making) (Burnes et al., 2023). RISE intervenes with the individual older adult OAM victim and alleged harmer (when appropriate), their relationship, and strengthens their informal and formal social supports.
  Arms: RISE-APS
Behavioral: APS — APS focuses on three main phases: case intake, investigation/ assessment, and substantiation/determination.

SUMMARY:
The goal of this study is to learn if the intervention, RISE (in partnership with APS), can be implemented in different contexts and if this RISE-APS model works in supporting older adults who are at risk of or experiencing some form of elder abuse or self-neglect. The main aims are to:

1. Adapt and implement the RISE-APS model in four new contexts
2. Evaluate the RISE-APS model implementation and effectiveness in four new locations

Researchers will compare outcomes of participants who receive APS-only services to those receiving the RISE-APS model to see if the RISE-APS model works better in supporting older adults.

Participants will:

Receive services in either group and participate in brief telephone surveys to track their outcomes over time.

DETAILED DESCRIPTION:
Elder abuse and self-neglect (EASN) are recognized by researchers, clinicians, and policymakers as pervasive problems with serious consequences for the aging population. EA is defined as an intentional act or lack of action by a person in a relationship involving an expectation of trust causing harm or risk of harm to an older adult; it comprises abuse (emotional/psychological, physical, sexual), neglect, and financial exploitation. SN, closely associated with EA, refers to the failure or inability of a person to satisfy their basic needs and protect themselves from harm. About 10% to 29% of community-dwelling older adults in the U.S. experience EASN each year. EASN is associated with serious consequences, such as premature mortality, poor physical and mental health, increased healthcare costs and utilization, and nursing home placement.

Without effective prevention and intervention strategies, the absolute scope of EASN will expand with the growth in the older adult population. In turn, community based EASN response programs, such as Adult Protective Services (APS), are under increasing pressure to address rising numbers of EASN case referrals and victims' need for support. Despite an increasing volume of case referrals, our understanding of effective EASN interventions represents a major gap in the field. Systematic reviews routinely find that the quality of EASN intervention research is weak and, in turn, strength of evidence is limited.

APS is the primary public agency responsible for receiving and responding to reports of EASN in the U.S. The current APS practice model typically focuses on three main phases: case intake, investigation/ assessment, and substantiation/determination. In 2021, at intake, APS received about 1.35 million reports of maltreatment allegations, and it accepted almost 797,000 cases for investigation. Among investigated cases, nearly 269,000 cases were substantiated. Although some APS programs provide services/referrals to address immediate client safety needs during and/or following the investigation phase, generally APS systems lack a dedicated, defined, and evidenced-based intervention phase to address underlying needs and risk factors. ACL guidelines recommend that effective APS models include a distinct service planning and intervention phase.

RISE (Repair Harm, Inspire Change, Support Connection, Empower Choice) was developed to address this intervention service gap in the APS EASN response system, based on prior research, theory, consultations with older adults and key stakeholders, and pilot testing. It was designed to address challenges that historically have limited EASN intervention capacity to address underlying case needs and risks, strengthen social supports, fulfill client priorities, and achieve more sustainable, holistic outcomes. RISE is informed by an ecological-systems intervention perspective, suggesting that effective models of EA intervention should have the capacity to work with both older adult victims and alleged harmers, their relationships, as well as to strengthen social supports surrounding them to address the full scope of risk factors that characterize a case. RISE is also informed by a person-centered practice orientation grounded in principles of client self-determination, cultural humility, and relationship building. RISE operates at Relational, Individual, Social, and Environmental levels of ecological influence and its core modalities seek to Repair Harm (restorative approaches), Inspire Change (motivational interviewing), Support Connection (teaming), and Empower Choice (supported decision-making).

Under the RISE-APS model, APS workers refer clients to RISE (with their consent). RISE "advocates" implement the intervention, engaging and building relationships with the victim, (and if they want, the harmer or others, or on their relationships) and working collaboratively with one or more of them. Advocates receive training in and employ specific core modalities that define the RISE model. Motivational interviewing, which has shown evidence to reduce EA re-victimization risk and advance intervention goals, is used to help victims and harmers resolve ambivalence and elicit openness to the change process . Teaming is employed to engage both informal and formal supports to surround the victim (and others if wanted), leveraging the known protective mechanisms of social support in EA cases (MacNeil et al., 2022). Restorative approaches are used with victims, alleged harmers, and others to help repair harm, hold harmers accountable and, where appropriate, restore relationships. Given the importance of the client-practitioner relationship in facilitating successful case outcomes, advocates are trained in engagement skills to navigate this threshold phase. RISE model core modalities described above were selected in part because they foster client-practitioner engagement and stronger relationships. To help facilitate behavioral change, goal setting is used as a dynamic process throughout the RISE intervention using a collaborative strategy called Goal Attainment Scaling, which has shown feasibility with APS clients.

RISE advocates deliver the intervention in person, over the phone, or using virtual teleconferencing methods, depending on client preference and safety needs. Interactions involve talk-based forms of support. Cases remain open, on average, approximately 5 months across phases of engagement, action, monitoring, and closure and involve sessions approximately 1-2 times/week. Similar to other EASN response programs, it is not possible to provide standardized information regarding the number and frequency of sessions or interactions with each case. EASN cases are highly heterogenous with varying needs, and outcomes of success across cases are multifarious. Cases are different in regard to mistreatment type(s) (or presenting issue), urgency and problem severity, circumstances and needs, perpetrator relationship and dynamics, and a host of other factors. Given the highly contextualized nature of EA cases, the number and frequency of RISE sessions vary across cases.

Beginning as a pilot in two randomly selected Maine counties in 2019 in partnership with APS, the RISE-APS model has since been scaled throughout the entire state. The RISE-APS ((R)epair Harm, (I)nspire Change, (S)upport Connection, €mpower Choice - Adult Protective Services) model has demonstrated evidence of feasibility, acceptability, and improvement in case outcomes (efficacy) in Maine, where RISE and APS have established a successful, complimentary partnership and referral process involving over 1500 cases to date. Among active clients, 77% have reported that RISE met most or almost all of their needs, and 89% reported being mostly or very satisfied with program services. In qualitative interviews, Maine APS caseworkers who refer cases to and work directly with RISE describe the partnership as collaborative and as integrating complimentary services; they also commonly report that RISE contributes to their own psycho-emotional well-being. Cases receiving the RISE-APS model in Maine significantly showed a 55% lower likelihood of re-investigation (recidivism) back in the APS system compared to cases receiving APS service alone. This protective effect of the RISE-APS model applied to nearly all forms and combinations of EASN. These findings suggested that both RISE and APS play critical, complementary roles in Maine within the overall EASN prevention/response system and that the combination of RISE-APS services appears to be most effective.

Goals and Objectives

Research shows initial evidence for the RISE-APS model in Maine. Further work is required to understand whether the RISE-APS model works in other contexts. Research is required to test the adaptation, implementation, and effectiveness of the RISE-APS model in different locations that serve older adults and families from varying communities. Addressing this need, this study will test the adaptation and effectiveness of the RISE-APS model in three new locations that each involve an APS program (making referrals to RISE) and a non-profit organization (housing and administering RISE): Ventura County, California (Ventura County APS, ONEgeneration); Harris County, Texas (Harris County APS, Harris County Area Agency on Aging), West Central, Texas (Northwest District APS, West Central AAA), and Cuyahoga County, Ohio (Cuyahoga County APS, Benjamin Rose). This study contains the following objectives and phases:

1. Adapt and implement the RISE-APS model in three new contexts
2. Evaluate the RISE-APS model implementation and effectiveness in three new locations

ELIGIBILITY:
Inclusion Criteria:

* APS cases assigned for investigation involving older adults age 60 years or older who live in the community and APS has assessed as at risk of or experiencing some form of elder abuse or self-neglect

Exclusion Criteria:

* APS clients who refuse services or who live in long-term care settings

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of Adult Protective Services Re-Investigations | Six months
  Number of Adult Protective Services (APS) re-investigation will be measured as the number of repeat APS investigations opened on a client in the 6 months following initial case closure during the study period
Adult Protective Services Re-Victimization | 6 months
  Adult Protective Services (APS) re-victimization will be measured as whether or not a client is determined to have experienced a substantiated maltreatment allegation at APS within 6 months following initial case closure during the study period.

SECONDARY OUTCOMES:
PROMIS Emotional Support | 4 months: Two data collection times (pre/post) at beginning of intervention (T0) and four-month post (T2)
  Emotional support will be measured using four items from the Patient-Reported Outcomes Measurement Information System (PROMIS) toolbox and assessed with response options from 0 (Never) to 4 (Always).
Number of Days to Adult Protective Services Re-Investigation | 6 months
  Number of days to adult protective services (APS) re-investigation will be measured as the number of days between initial case closure and when a case is reopened for investigation at APS within a 6 month period.
PROMIS General Self-Efficacy | 4 months: Two data collection times (pre/post) at beginning of intervention (T0) and four-month post (T2)
  General Self-Efficacy will be measured using four items from the Patient-Reported Outcomes Measurement Information System (PROMIS) toolbox and assessed with response options from 0 (Never) to 4 (Always).
PROMIS Perceived Stress | 4 months: Two data collection times (pre/post) at beginning of intervention (T0) and four-month post (T2)
  Perceived stress will be measured using four items from the Patient-Reported Outcomes Measurement Information System (PROMIS) toolbox and assessed with response options from 0 (Never) to 4 (Always).
RISE Intervention Client Adoption | 2 years
  RISE intervention client adoption will be measured by the proportion of eligible clients who are referred to RISE and accept services

OTHER OUTCOMES:
RISE Intervention Adoption by Adult Protective Services Caseworkers | 2 years
  RISE intervention adoption will be measured by the proportion of APS caseworkers referring to RISE

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - ONEgeneration and Ventura County APS, Reseda, California
  - Benjamin Rose and Cuyahoga County APS, Cleveland, Ohio
  - Area Agency on Aging of West Central Texas; Northwest District APS, Abilene, Texas
  - Harris County APS and Area Agency on Aging, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Older adult elder abuse victim participant recruitment into this study is very challenging, including participation in pre/post participant surveys to collect primary outcomes. Sharing data with other researchers may restrict our capacity to recruit this already challenging community of prospective participants.

REFERENCES:
- [Background] Burnes D, MacNeil A, Connolly MT, Salvo E, Kimball PF, Rogers G, Lewis S. A qualitative evaluation of the "RISE" elder abuse intervention from the perspective of adult protective services caseworkers: addressing a service system gap. J Elder Abuse Negl. 2022 Nov-Dec;34(5):329-348. doi: 10.1080/08946566.2022.2140321. Epub 2022 Oct 31. PMID 36316963
- [Background] AMH completes transition to important functions. Jt Comm Perspect. 1994 May-Jun;14(3):1, 7-8. No abstract available. PMID 10136376
- [Background] Ooie T, Saikawa T, Hara M, Ono H, Seike M, Sakata T. H2-blocker modulates heart rate variability. Heart Vessels. 1999;14(3):137-42. doi: 10.1007/BF02482297. PMID 10776806
- [Background] Saadia R, Schein M. Multiple organ failure. How valid is the "two hit" model? J Accid Emerg Med. 1999 May;16(3):163-6; discussion 166-7. doi: 10.1136/emj.16.3.163. PMID 10353038
- [Background] Moussaoui F, Michelutti I, Le Roux Y, Laurent F. Mechanisms involved in milk endogenous proteolysis induced by a lipopolysaccharide experimental mastitis. J Dairy Sci. 2002 Oct;85(10):2562-70. doi: 10.3168/jds.S0022-0302(02)74339-7. PMID 12416808
- See also: Intervention website — https://risecollab.org/